CLINICAL TRIAL: NCT06890000
Title: Effectiveness of Scapular Exercises Compared To Conventional Treatment in People With Shoulder Pain: A Randomized Controlled Study
Brief Title: Effectiveness of Scapular Exercises Compared To Conventional Treatment in Shoulder Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mehmet Delen, Asst Prof, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09/972
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Pain; Scapular Dyskinesis
Keywords: Shoulder pain; obvious scapular dyskinesis; Conventional Treatment; Scapular Exercises; Effectiveness
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Scapular Exercises (Experimental): Scapular exercise includes scapular clock exercise, rowing exercise, resisted external rotation, resisted punching exercise.
  The group program also includes conventional treatment.
  Interventions: Other: Scapular Exercise; Other: Control (Standard treatment)
- Conventional Treatment (Active Comparator): Conventional treatment includes TENS, hotpack, Stretching exercises (posterior capsule and pectoral muscle), resisted flexion and abduction exercises
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Scapular Exercise — Scapular exercise includes scapular clock exercise (3 sets of 10 repetitions), rowing exercise (3 sets of 10 repetitions), resisted external rotation (3 sets of 10 repetitions), resisted punching exercise (3 sets of 10 repetitions).
  The rowing, external rotation and punching exercises will do with theraband. When participants complete the elastic band exercises easily and do not report any muscle fatigue, they will move on to the next level of difficulty. The color order of the bands is yellow, red, green and blue. The exercises will begin with the yellow elastic band, which provides the least resistance.
  The intervention will last for 6 weeks, with 2 training sessions per week and each training session lasting 15-20 minutes.
  Arms: Scapular Exercises
Other: Control (Standard treatment) — Conventional Treatment includes TENS (100 Hz) with hotpack (20 minutes), Stretching exercises (posterior capsule and pectoral muscle), resisted flexion and abduction exercises.
  The rowing, external rotation and punching exercises will do with theraband. When participants complete the elastic band exercises easily and do not report any muscle fatigue, they will move on to the next level of difficulty. The color order of the bands is yellow, red, green and blue. The exercises will begin with the yellow elastic band, which provides the least resistance.
  The intervention will last for 6 weeks, with 2 training sessions per week and each training session lasting 30-45 minutes.

SUMMARY:
The contribution of the scapula to shoulder joint movement is great. The contribution of the scapula bone is more prominent, especially in overhead activities. Therefore, the position and movement of the scapula are generally examined in people with shoulder disease. Scapula-focused exercises are used in patients with shoulder problems. However, some studies focused on the effectiveness of scapula-focused exercises on shoulder problems. Thes studies fundings are controversial. Scapular dyskinesis has not been evaluated in these studies. No study has set the condition of having scapular dyskinesis as an inclusion criterion. Scapular-focused exercises are expected to have a greater effect especially on patients with scapular dyskinesis. Therefore, the aim of this study is to examine the effectiveness of scapula-focused exercises on patients with shoulder pain and obvious scapular dyskinesis.

ELIGIBILITY:
Inclusion Criteria:

* Having shoulder pain for at least 1 month
* Having obvious scapular dyskinesia
* Having a shoulder ROM (range of motion) at least 120º
* Being 18 years of age or older

Exclusion Criteria:

* Having received any shoulder treatment in the last 6 months
* Having an acromioclavicular joint problem
* Having a diagnosis of frozen shoulder
* Having a fracture in the shoulder area
* Having a major rotator cuff muscle tear
* Having a diagnosis of calcific rotator cuff tendinopathy
* Having a neurological or rheumatological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
shoulder pain and disability index (SPADI) | Baseline and at 6 week
  SPADI is a self reported outcome for shoulder disorders. SPADI includes 13 questions. Scores range from 0 to 100. The higher a patient scores on the SPADI, the greater the level of pain/disability.

SECONDARY OUTCOMES:
Global Rate of Change | Baseline and at 6 week
  GRoC is a reliable assessment method with 11 levels, frequently used to track changes in a participant's condition. Participants who selected the top two categories (much better and very much better) were considered recovered.

CONTACTS AND LOCATIONS:
Locations (1):
- Universtiy of Health Sciences - Gülhane Faculty of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to data protection rules

REFERENCES:
- [Background] Bury J, West M, Chamorro-Moriana G, Littlewood C. Effectiveness of scapula-focused approaches in patients with rotator cuff related shoulder pain: A systematic review and meta-analysis. Man Ther. 2016 Sep;25:35-42. doi: 10.1016/j.math.2016.05.337. Epub 2016 Jun 4. PMID 27422595